CLINICAL TRIAL: NCT01717001
Title: In Vivo Determination & Comparison of Knee Kinematics for Subjects Implanted With Either a Personalized ConforMIS or Traditional Knee Implant
Brief Title: Comparison of Knee Kinematics for Subjects Implanted With Either a ConforMIS or Traditional Knee Implant
Status: Completed | Type: Observational
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Other Study IDs: Komistek 1
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Results first posted 2020-12-31 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
Keywords: kinematics; knee joint
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ConforMIS: Patients with ConforMIS implants
- Standard Total Knee Implant: Patients implanted with standard total knee implant

SUMMARY:
A better understanding of knee joint kinematics is important to explain the premature polyethylene wear failures within total knee arthroplasties (TKAs) and to help design a prosthesis that most closely approximates the normal knee. Previously, most experimental studies of knee kinematics have involved cadaveric, in vitro analyses, or have not tested the knee in a weight-bearing mode. Others have used exoskeletal linkages and skin markers that permit error due to undesired motions between markers and the underlying bone. More recently, fluoroscopy has been used to assess in vivo kinematics for subjects having a TKA.

ConforMIS has attempted to follow a clearly different path than the major orthopaedic companies. They have chosen to offer patients a personalized knee implant based off of each patient's femoral and tibial bone geometry. The hypothesis is that these subjects will experience a more normal-like kinematic pattern, eliminating paradoxical anterior sliding during weight-bearing knee flexion. Therefore, the objective for this study is to analyze the in vivo kinematics for 25 patients implanted with a personalized ConforMIS TKA and 25 patients implanted with a traditional TKA design to determine if there are any kinematic differences between these TKA designs.

DETAILED DESCRIPTION:
Each subject will be asked to perform five activities in one continuous sequence: (1) stand up from a chair, (2) walk up stairs, (3) walk down stairs, (4) level walking, and (5) a deep knee bend. Subjects will be video recorded from the waist down while performing the activities. The speed level of each trial will be based on the comfort level of the patient. The fluoroscopic images will be stored digitally for subsequent analysis on secure servers and workstations at the University of Tennessee.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months post-op with no other surgical procedures conducted within the past 6 months
* Between 40-70 years of age
* Body weight of less than 250lbs
* BMI of less than 38
* Pregnant females will be excluded
* TKA patients will be judged Clinically successful with an American Knee Society score of greater than 90
* Must have 100 degrees post-op passive flexion with no ligamentous laxity or pain
* Participants must be able to walk on level ground without aid of any kind and ascend/descend stairs without assistance.
* All potential subjects will have either a personalized ConforMIS™ TKA or a traditional TKA manufactured by an orthopaedic company other than ConforMIS.
* Patients from the physician's list who do not meet the study requirements will not be considered.
* Patients must be willing to sign the Informed Consent and HIPAA forms to participate in the study.
* Patients must be between 160cm (5'3) and 193cm (6'4) tall.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 6 month post-op with a ConforMIS knee replacement or a standard total knee replacement who meets the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Komistek, PhD, Principal Investigator — Univeristy of Tennessee; William Kurtz, MD, Principal Investigator — Tennessee Orthopedic Alliance
Locations (2):
- United States (2):
  - University of Tennessee, Knoxville, Tennessee
  - Tennessee Orthopedic Alliance, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ConforMIS | Standard Total Knee Implant
Started | 38 | 28
Completed | 32 | 24
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Population: Subjects who were implanted with either a first generation iTotal CR (Conformis arm) or PS (Standard Total Knee Implant arm) were not included in analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | ConforMIS | Standard Total Knee Implant | Total
Number analyzed (Participants) | 24 | 14 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (7.7) | 66.7 (5.7) | 62.6 (7.6)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data not accessible and not used for analysis Population: Data not accessible and not used for analysis
Region of Enrollment [Number; unit: participants]
  United States | 24 | 14 | 38

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Range of Motion
Description: Comparison of amount of flexion achieved by the knee between the two arms
Time Frame: at least 6 months post-surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | ConforMIS | Standard Total Knee Implant
Number analyzed (Participants) | 24 | 14
degrees | 103.8 (14.7) | 95.8 (21.2)

ADVERSE EVENTS:
Arm/Group | ConforMIS | Standard Total Knee Implant
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/14
Other Adverse Events (participants affected / at risk) | 0/24 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No